CLINICAL TRIAL: NCT04308525
Title: Optimising Microsurgical Reconstruction After Advanced Head and Neck Cancers - Enhanced Recovery and Improved Clinical Pathway
Brief Title: Optimising Microsurgical Reconstruction After Advanced Head and Neck Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Hjermind Højvig, M.D., Ph.D.-student, Rigshospitalet, Denmark
Other Study IDs: ERAS Free FLAP for H&N Cancer
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: free flap; microsurgery; microvascular reconstruction; Enhanced recovery after surgery; ERAS
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Early Ambulation; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS Group: Prospectively included patients after introduction of an ERAS programme
  Interventions: Behavioral: Early ambulation; Behavioral: Early oral feeding; Other: Multimodal opioid-sparing analgesia; Procedure: Goal-directed fluid therapy; Procedure: CAD/CAM system for reconstructive plates; Other: Functional discharge criteria
- Control group: We retrospectively evaluated our procedures for the period 2014-2016
  Interventions: Other: Standard/historical postoperative regimen

INTERVENTIONS:
Behavioral: Early ambulation — Early ambulation will help prevent postoperative infections, especially pneumonia and urinary tract infections. Additionally it will prevent constipation by promotion of bowel-movement and function and prevent thromboembolic complications. Patients undergoing surgery with a free fibula flap are currently unable to ambulate for 6 to 7 days while a split-thickness skin-graft is healing. We will apply a pressure dressing to the wound which makes ambulation possible immediately after surgery (or after return from the ICU). Likewise, all other patient groups will be encouraged to fully ambulate on POD (post-operative day) 1 or POD 2.
  Groups: ERAS Group
Behavioral: Early oral feeding — To monitor the patients' nutritional status, blood samples will be taken to identify risk of refeeding syndrome and patients will be evaluated according to the current guidelines from the ENT (ear-, nose-, throat-) department. We wil use the ESPEN guidelines for nutritional risk screening (NRS-2002), which have been validated for head and neck cancer patients to perform a risk assessment for malnutrition. A consultation with a clinical dietician will be arranged in order to calculate the required daily nutritional intake. Patients in risk of refeeding syndrome will be closely monitored in the outpatient clinic during the time from the MDT(Multi Disciplinary Team) conference to the day of surgery. Patients in need of additional nutritional support will be provided with supplementary energy/protein drinks. Some patients may need closer monitoring, guidance regarding extra meals and to have a nasogastric tube placed to get used to the tube and optimize pre-operative nutritional status.
  Other Names: Focus on nutritional status
  Groups: ERAS Group
Other: Multimodal opioid-sparing analgesia — On-label use of already approved drugs including perioperative dexamethasone, administered with the aim of reducing opioid intake.
  Pre-operatively the patients are given 400 mg of Celebra. During surgery 24 mg of dexamethasone is administered. The post-operative regimen consists of 12 mg of Dexamethasone 48 and 96 hours post-operatively, 200 mg of Celebra morning and evening (maximum 14 days) and 1g of paracetamol times four times daily. Morphine will only be administered when assessed necessary with a dose of 10 mg p.n. maximum six times a day.
  Groups: ERAS Group
Procedure: Goal-directed fluid therapy — Focus on avoidance of over-hydration. Aim for fluid-load after surgery: max: +1000-1500 ml
  Groups: ERAS Group
Procedure: CAD/CAM system for reconstructive plates — Computer-assisted design and modelling (CAD/CAM) are a system for pre-operative planning and construction of reconstructive plates used for mandibular reconstruction. This will help reduce the operating-time, as the maxillofacial surgeon will bring a pre-bent reconstructive plate to the procedure instead of manually forming it during surgery. Already implemented for several procedures in the department.
  Other Names: Minimally invasive surgery
  Groups: ERAS Group
Other: Functional discharge criteria — Introduction of a number of functional discharge criteria to avoid prolonged postoperative hospitalisation
  Groups: ERAS Group
Other: Standard/historical postoperative regimen — Non-formalised historical peri- and postoperative regimen.
  Groups: Control group

SUMMARY:
This study aims to improve the peri- and postoperative care regimen for patients undergoing microvascular reconstruction after head and neck cancer by introducing an enhanced recovery after surgery (ERAS) programme.

DETAILED DESCRIPTION:
Advanced stage head and neck cancers have a poor prognosis and a 5-year survival rate of as low as 35-37%. The treatment is complex and often requires a multidisciplinary approach including surgery. The goal besides removal of the cancer is to restore function and appearance. If possible, both resection as well as immediate reconstruction will be performed during the same surgical procedure. Due to the large bone- and soft tissue loss following the ablative procedure, local solutions are often inadequate for reconstruction. In addition, many patients require post-operative radiotherapy, which may result in tightness of scar tissue and impaired function. In these cases it is necessary to perform the reconstruction using a free flap.

Free flap reconstruction involves tissue taken from other parts of the body, that is transplanted along with the associated blood vessels to the reconstruction site. The vessels of the flap are usually anastomosed to the vessels of the neck (microvascular reconstruction) and the transplanted tissue thereby obtains a blood supply at its new location. Head and neck cancer patients are usually reconstructed using the free fibular flap, the latissimus dorsi flap, the radial forearm flap or the anterolateral thigh flap.

The combination of complicated surgery and often malnourished patients with a low body mass index (BMI), that typically suffer from tobacco and alcohol abuse, commonly lead to postoperative ICU treatment and complications. The most common are infections, re-operations, delayed wound healing and refeeding syndrome, which is reported in up to 35% of patients undergoing major surgery for head and neck cancer.

Even with successful reconstruction, many patients suffer from drooling, lack of adequate clenching, permanent gastric tube feeding, insufficient wound healing and a high recurrence rate. Enhanced recovery after surgery (ERAS) is a peri- and postoperative care concept designed to accelerate recovery and improve convalescence. It has previously been established as superior to conventional care for a wide variety of procedures. As one of the first departments in the world our department has successfully implemented an ERAS program for microsurgical patients that undergo breast reconstruction using autologous tissue. By utilizing our experience with ERAS and combining it with a review of our own patient data we have developed an ERAS protocol for microvascular reconstruction after ablative surgery for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for ablative surgery for head and neck cancer with primary microvascular reconstruction.

Exclusion Criteria:

* Patients with conditions leading to increased risk of thromboembolic events
* Patients pre-operatively admitted to the ICU

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery and microvascular reconstruction for head and neck cancers. Procedures may be "primary" or for recurrent disease.
  Patients often suffer from several comorbidities. Most patients have a history of tobacco use. Prognosis is poor and five-year rate of survival is 35-37%.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay (LOS) | 1 to 4 weeks
  Time from surgery to discharge

SECONDARY OUTCOMES:
ICU LOS | 1-2 days
  Time spent in the ICU (intensive care unit) post-operatively
Time to ambulation | 1-7 days
  Days from surgery until full ambulation (walking)
Incidence of infections | 30 days
  Number of postoperative infections
Incidence of re-operations | 30 days
  Number of return-to-theatre events
Complication-rate | 30 days
  Number of surgical related complications

CONTACTS AND LOCATIONS:
Overall Officials: Jens H Hojvig, Md, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, København Ø, Denmark

REFERENCES:
- [Background] Hanasono MM, Friel MT, Klem C, Hsu PW, Robb GL, Weber RS, Roberts DB, Chang DW. Impact of reconstructive microsurgery in patients with advanced oral cavity cancers. Head Neck. 2009 Oct;31(10):1289-96. doi: 10.1002/hed.21100. PMID 19373778
- [Background] Montero PH, Patel SG. Cancer of the oral cavity. Surg Oncol Clin N Am. 2015 Jul;24(3):491-508. doi: 10.1016/j.soc.2015.03.006. Epub 2015 Apr 15. PMID 25979396
- [Background] Bak M, Jacobson AS, Buchbinder D, Urken ML. Contemporary reconstruction of the mandible. Oral Oncol. 2010 Feb;46(2):71-6. doi: 10.1016/j.oraloncology.2009.11.006. Epub 2009 Dec 29. PMID 20036611
- [Background] Wei FC, Chen HC, Chuang CC, Noordhoff MS. Fibular osteoseptocutaneous flap: anatomic study and clinical application. Plast Reconstr Surg. 1986 Aug;78(2):191-200. doi: 10.1097/00006534-198608000-00008. PMID 3523559
- [Background] Omura K. Current status of oral cancer treatment strategies: surgical treatments for oral squamous cell carcinoma. Int J Clin Oncol. 2014;19(3):423-30. doi: 10.1007/s10147-014-0689-z. Epub 2014 Apr 1. PMID 24682763
- [Background] Rasmussen SO, Kristensen MB, Wessel I, Andersen JR. Incidence and Risk Factors of Refeeding Syndrome in Head and Neck Cancer Patients-An Observational Study. Nutr Cancer. 2016 Nov-Dec;68(8):1320-1329. doi: 10.1080/01635581.2016.1225103. Epub 2016 Sep 28. PMID 27682582
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Bonde CT, Khorasani H, Elberg J, Kehlet H. Perioperative Optimization of Autologous Breast Reconstruction. Plast Reconstr Surg. 2016 Feb;137(2):411-414. doi: 10.1097/01.prs.0000475749.40838.85. PMID 26818274